CLINICAL TRIAL: NCT02069847
Title: Prospective Evaluation of the Clinical Utility of Budesonide for the Prevention of Esophageal Strictures After Endotherapy
Brief Title: Prospective Evaluation of Budesonide for Prevention of Esophageal Strictures After Endotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Wallace, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-009467
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Stricture
Keywords: Esophageal stricture formation; Endoscopic mucosal resection; Endoscopic submucosal dissection; Budesonide; Radical endoscopic mucosal resection; EMR; ESD
MeSH Terms: conditions — Esophageal Stenosis | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esophageal stricture, Budesonide (Experimental): Budesonide 1mg twice a day for a total of 8 weeks following endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR)
  Interventions: Drug: Budesonide
- Control group (No Intervention): Retrospective collect data for subjects who undergo endoscopic submucosal dissection or endoscopic mucosal resection

INTERVENTIONS:
Drug: Budesonide — Participants will be instructed to swallow budesonide 3mg twice daily for eight consecutive weeks following endotherapy with EMR or ESD. Budesonide will be provided in a capsule containing 3mg budesonide only by Mayo Clinic Pharmacy with full 8 weeks supply.
  The patient will require opening the capsule and mixing the budesonide powder in 10ml (2 teaspoons) honey, or pancake syrup.
  Patients will be instructed not to ingest any solid or liquids for 30 minutes before and after taking the budesonide. For purposes of this study, budesonide is used off-label but according to the same dose and efficacy as has been demonstrated in other esophageal inflammatory conditions. Patients will receive a handout with exact instructions how and when to take Budesonide.
  Other Names: Budesonide, Entocort, Uceris
  Arms: Esophageal stricture, Budesonide

SUMMARY:
Surgery has been historically the mainstay treatment for advanced pre-malignant lesions and early esophageal cancers. However, esophagectomy is associated with significant morbidity and mortality. With the advance of therapeutic endoscopy, there has been a growing interest and application of endoscopic resection and mucosal ablative techniques for the treatment of these diseases. Esophageal stricture (ES) formation has become an increasingly recognized complication of extensive endoscopic mucosal ablation and/or resection. The resultant symptomatic stricture development can significantly impair a patient's quality of life. Endoscopic therapy of esophageal strictures with balloon dilation and/or local steroid injection is invasive, costly, and associated with the potential risk of perforation. Recently, oral corticosteroids have been introduced for the prevention of esophageal stricture after endoscopic submucosal dissection.

Budesonide is a synthetic steroid with topical anti-inflammatory properties and high first-pass metabolism; thus, potentially less systemic absorption and side effects.

Hypothesis: Oral budesonide prevents esophageal stricture formation in patients who underwent radical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) for advanced premalignant esophageal lesions or superficial esophageal cancers.

DETAILED DESCRIPTION:
Esophageal stricture (ES) formation is a widely recognized adverse event of radical EMR and ESD. Indeed, ES is the most common complication of radiofrequency ablation (RFA) for Barrett's esophagus (BE), with a reported incidence ranging from 5% to 12%. A single-center retrospective study reported ES formation in 67% of 73 patients with EMR of at least 50% of their esophageal circumference. Similarly, the incidence of ES development after ESD is between 70-90% when the mucosal defect involves more than three-quarters of the esophageal circumference. In aggregate, the extent of the esophageal mucosal defect following endotherapy appears to be the most consistent predictor of ES formation. Prevention of ES development following endotherapy can significantly improve a patient's quality of life and possibly reduce the potential risks and costs associated with treatment of ES with repeated endoscopic balloon dilations (EBD). Glucocorticoids have been evaluated as a potential preventive therapy for ES based on their anti-inflammatory properties and inhibitory effects on collagen deposition. Oral prednisolone has been shown to be effective as a preventive strategy for ES formation. However, prolonged use of systemic oral steroids can be associated with multiple adverse effects.

Budesonide is a synthetic steroid with topical anti-inflammatory properties and high first-pass metabolism; thus, potentially less systemic absorption and side effects. Most recently Mayo Clinic Rochester developed a new budesonide capsule formulation. Alike viscous budesonide the budesonide capsule can be opened and the powder can be mixed with honey or pancake syrup. A similar formulation is currently used in pilot studies for treatment of eosinophilic esophagitis. The advantage of budesonide capsule is the improve taste in comparison to viscous budesonide originating from budesonide respules which is unpalatable.

Study aims:

1. The aim of this study is to prospectively record our experience with budesonide for the prevention of esophageal stricture formation after endotherapy (mucosal resection, submucosal dissection) as part of routine medical care.
2. The data will be compared with outcomes with well-annotated historical controls that underwent similar procedure with similar follow up but without budesonide exposure.
3. If sufficient efficacy is seen, these data will be used to plan a prospective controlled clinical trial. All patients in the study group will receive standard medical care and no experimental interventions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of esophageal lesion treated with ESD or EMR which involves ≥ 50% of the esophageal circumference.

Exclusion Criteria:

* Locally advanced disease
* Prior esophageal surgery
* Participation in another research protocol that could interfere or influence the outcome measures of the present study.
* The subject or legal representative is unable/unwilling to give informed consent. (study group)
* Medications or conditions for which there is a contraindication to use of budesonide (see pharmacology section below)
* Concomitant use of systemic steroids or other immune suppressive medication for a different condition 9. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02; Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wallace, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Esophageal Stricture, Budesonide: Budesonide 1mg twice a day for a total of 8 weeks following endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR)
  Budesonide: Participants will be instructed to swallow budesonide 3mg twice daily for eight consecutive weeks following endotherapy with EMR or ESD. Budesonide will be provided in a capsule containing 3mg budesonide only by Mayo Clinic Pharmacy with full 8 weeks supply.
  The patient will require opening the capsule and mixing the budesonide powder in 10ml (2 teaspoons) honey, or pancake syrup.
  Patients will be instructed not to ingest any solid or liquids for 30 minutes before and after taking the budesonide. For purposes of this study, budesonide is used off-label but according to the same dose and efficacy as has been demonstrated in other esophageal inflammatory conditions. Patients will receive a handout with exact instructions how and when to take Budesonide.
Period: Overall Study
Arm/Group | Esophageal Stricture, Budesonide | Control Group
Started | 22 | 68
Completed | 22 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Esophageal Stricture, Budesonide: Budesonide 1mg twice a day for a total of 8 weeks following endoscopic submucosal dissection or endoscopic mucosal resection
  Budesonide: Participants will be instructed to swallow budesonide 3mg twice daily for eight consecutive weeks following endotherapy with EMR or ESD. Budesonide will be provided in a capsule containing 3mg budesonide only by Mayo Clinic Pharmacy with full 8 weeks supply.
  The patient will require opening the capsule and mixing the budesonide powder in 10ml (2 teaspoons) honey, or pancake syrup.
  Patients will be instructed not to ingest any solid or liquids for 30 minutes before and after taking the budesonide. For purposes of this study, budesonide is used off-label but according to the same dose and efficacy as has been demonstrated in other esophageal inflammatory conditions. Patients will receive a handout with exact instructions how and when to take Budesonide.
- Total: Total of all reporting groups
Arm/Group | Esophageal Stricture, Budesonide | Control Group | Total
Number analyzed (Participants) | 22 | 68 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (10.6) | 67.9 (10.3) | 70.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 18 | 58 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22 | 68 | 90

OUTCOME MEASURES:

1. Primary Outcome: Dysplasia in Barrett Esophagus (BE)
Description: Number of subjects with Non-dysplastic, low grade dysplasia, high grade dysplasia and T1a early esophageal adenocarcinoma. As measured by using the BE dysplasia grading system of Non-dysplastic (no cancerous tissue present), low-grade dysplasia (minor cell changes found), high-grade dysplasia (extensive cell changes found, but not yet cancer), and noninvasive cancer (T1a early esophageal adenocarcinoma)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Stricture, Budesonide | Control Group
Number analyzed (Participants) | 22 | 68
Participants
  Non-dysplastic BE | 4 | 4
  Low grade dysplasia BE | 3 | 23
  High grade dysplasia BE | 6 | 20
  T1a early esophageal adenocarcinoma | 9 | 20
Statistical Analysis 1: Comparison: Esophageal Stricture, Budesonide vs Control Group; Test type: Superiority; p = 0.992, ANOVA

2. Secondary Outcome: Rate of Esophageal Stricture
Description: Number of subjects with 50-74%, 75-99% and 100% esophageal stricture. Defined as the percentage of esophageal lumen narrowing requiring dilation prior to passage of the endoscope and/or presence of new dysphagia.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Stricture, Budesonide | Control Group
Number analyzed (Participants) | 22 | 68
Participants
  50-74% esophageal stricture | 1 | 9
  75-99% esophageal stricture | 0 | 6
  100% esophageal stricture | 3 | 0
Statistical Analysis 1: Comparison: Esophageal Stricture, Budesonide vs Control Group; Total number of budesonide subjects with 50% or greater esophageal stricture (N=4) vs total number of control subjects with 50% or greater esophageal structure (N=15); Test type: Superiority; p = 0.531, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were only collected on the prospective arm of the study, the Budesonide treatment arm and not available for the retrospective chart review of the control arm. Adverse events were collected for each subject from enrollment until 12 week follow up, for an overall study duration of approximately 3 years.
Arm/Group | Esophageal Stricture, Budesonide
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esophageal Stricture, Budesonide (N=22)
Dilation (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02069847/Prot_SAP_000.pdf